CLINICAL TRIAL: NCT01994187
Title: the Clinic Registration Study of Carotid Stenosis Revascularization
Brief Title: Revascularization of Extracranial Carotid Artery Stenosis
Acronym: RECAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XW125-S004
Record Dates: First submitted 2013-09-25; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Carotid Stenosis; Surgery; Stroke
Keywords: Carotid stenosis; Angioplasty; Carotid endarterectomy; Stroke
MeSH Terms: conditions — Carotid Stenosis; Stroke | interventions — Endarterectomy, Carotid; Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CAS or CEA: CAS:the patient who accepted carotid angioplasty due to catotid artery stenosis CEA:the patient who accepted carotid endarterectomy due to catotid artery stenosis
  Interventions: Procedure: Carotid endarterectomy; Procedure: carotid angioplasty

INTERVENTIONS:
Procedure: Carotid endarterectomy
  Other Names: conventional carotid endarterectomy; Eversion carotid endarterectomy
Procedure: carotid angioplasty
  Other Names: carotid angioplasty with stent

SUMMARY:
Investigate the current situation of carotid stenosis therapy in China. Establish the data bank of carotid stenosis revascularization (CAS and CEA) in China ,in order to get best quality control of the therapy, as well as confirm the standard treatment for carotid stenosis.

Understand situation about the adverse events occurs after the revascularization (CAS and CEA), evaluate the health economics .

DETAILED DESCRIPTION:
The carotid stenosis was one of the higher risk of the ischemia stroke in China.In the mean time ,more and more people accept revascularization because of carotid stenosis.NASCAT indicated that CEA is the "golden standard" of the therapy of the carotid stenosis.But in china , case the opposite,only little patient receive CEA,on the other hand , most patients received angioplasty.

Expected no less than 2100 cases within 2 years for the whole study. We choose 39 hospitals whose experienced in CAS or/and CEA spread all over the country as multiple centers for this clinic registration study. All cases inclusion must be continuously registration.

The subject choice:All registered patients must be signed informed consent to register for non intrusive research this study ,the researchers during the study period should be continuous registration in patients undergoing surgical treatment of carotid stenosis, to ensure that the selected participants reflect the target patient population.

Medical Center choice: This research for the study of the registration, therefore, when the choice, all the medical center will be based on market research data.

Primary endpoint or the main aim of this registration study is to observe the following details:

1. The participants who suffer from stroke(ischemic or hemorrhagic), death or cardiovascular events within 30 days after any revascularization procedure.
2. The participants who suffer from ipsilateral stroke(ischemic or hemorrhagic) or death beyond 30 days to 12 months after any revascularization procedure.

Secondary endpoint or the other aims of this registration study:

1. Success rate of any procedure (CAS or CEA).
2. postoperative complications, including hyperperfusion syndrome,TIA, ipsilateral infarction, vascular dissection and other adverse events.
3. To observe the rate of restenosis during follow-up.
4. Stroke in patients with TIA mainly heart attacks and other cardiovascular events during follow-up.
5. Changes of the patients with mRS NIHSS Barthel Index score.
6. Postoperative patients with drug use.
7. Patient survival after 12 months.
8. Patients hospitalized cost during follow-up.

This study does not need to be random. The study is expected to begin in July 2013 in the first, participants in the group stage for two years, to the end of June 2015 into the group of patients after surgery, follow-up of at least 12 months after the last case the participants into groups and followed up for 12 months, is expected to be completed in June 2015.

ELIGIBILITY:
Inclusion Criteria:all the consecutive cases of carotid stenosis which received CEA or/and CAS in central hospital during the study(upto 2015).

Exclusion Criteria:the cases of carotid stenosis which received CEA or/and CAS in other hospital(not enroll this study) will be exclusion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: one group:1050 cases of endarterectomy; the other group:1050 cases of carotid artery stent; totally:2100 cases of ravascularization for carotid stenosis
Sampling Method: Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The participants who suffer from stroke(ischemic or hemorrhagic), death or cardiovascular events within 30 days after any revascularization procedure. | 30 days
  The participants who suffer from stroke(ischemic or hemorrhagic), death or cardiovascular events within 30 days after any revascularization procedure.
The participants who suffer from ipsilateral stroke(ischemic or hemorrhagic) or death beyond 30 days to 12 months after any revascularization procedure. | beyond 30 days to 12 months
  The participants who suffer from ipsilateral stroke(ischemic or hemorrhagic) or death beyond 30 days to 12 months after any revascularization procedure.

SECONDARY OUTCOMES:
Success rate of any procedure (CAS or CEA) | 1 days
  Success rate of any procedure (CAS or CEA)
postoperative complications, including hyperperfusion syndrome,TIA, ipsilateral infarction, vascular dissection and other adverse events. | 7 days
  postoperative complications, including hyperperfusion syndrome,TIA, ipsilateral infarction, vascular dissection and other adverse events.
To observe the rate of restenosis during follow-up. | 12 months
  To observe the rate of restenosis during follow-up.
Stroke in patients with TIA mainly heart attacks and other cardiovascular events during follow-up. | 12 months
  Stroke in patients with TIA mainly heart attacks and other cardiovascular events during follow-up.
Changes of the patients with mRS NIHSS Barthel Index score | 12 months
  Changes of the patients with mRS NIHSS Barthel Index score
Postoperative patients with drug use | 12 months
  Postoperative patients with drug use
Patient survival after 12 months | 12 months
  Patient survival after 12 months
Patients hospitalized cost | 5-7 days
  Patients hospitalized cost

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ling, MD, Principal Investigator — Xuanwu Hospital, Capital University of Medical Sciences, Beijing, China
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, China

REFERENCES:
- [Derived] Yang B, Ma Y, Wang T, Chen Y, Wang Y, Zhao Z, Chen D, Wang J, Xu X, Luo T, Hua Y, Ling F, Qureshi AI, Hong B, Jiao L; RECAS Trial Investigators. Carotid Endarterectomy and Stenting in a Chinese Population: Safety Outcome of the Revascularization of Extracranial Carotid Artery Stenosis Trial. Transl Stroke Res. 2021 Apr;12(2):239-247. doi: 10.1007/s12975-020-00835-8. Epub 2020 Jul 19. PMID 32686047